CLINICAL TRIAL: NCT02776514
Title: Intraarticular Injections of Steroids, Hyaluronic Acid or Platelet Rich Plasma Versus Placebo for the Knee Osteoarthritis
Brief Title: Steroids, Hyaluronic Acid or Platelet Rich Plasma Versus Placebo for the Knee Osteoarthritis
Acronym: KIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Collaborators: Stiftung für Rheumaforschung Zurich (Unknown); Stiftung Marie-Lou Ringgenberg Bern (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W-560
Record Dates: First submitted 2016-02-18; First posted 2016-05-18 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Triamcort (1 ml, 40 mg/ml) (Active Comparator): 30 patients receive intraarticular injection with steroids (and contrast media Iopamiro 200)
  Interventions: Drug: Triamcort
- Platelet-rich-plasma (PRP 3 ml) (Active Comparator): 30 patients receive intraarticular injection with platelet-rich-plasma (PRP) (and contrast media Iopamiro 200)
  Interventions: Drug: Platelet-rich-plasma
- Suplasyn1-shot (60 mg/ ml) (Active Comparator): 30 patients receive intraarticular injection with hyaluronic acid (and contrast media Iopamiro 200)
  Interventions: Drug: Suplasyn1
- Placebo (Iopamiro 200) (Placebo Comparator): 30 patients receive intraarticular injection with contrast media only
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Triamcort — Fluoroscopic guided injection in the knee joint
  Arms: Triamcort (1 ml, 40 mg/ml)
Drug: Platelet-rich-plasma
  Arms: Platelet-rich-plasma (PRP 3 ml)
Drug: Suplasyn1
  Arms: Suplasyn1-shot (60 mg/ ml)
Drug: Placebo
  Arms: Placebo (Iopamiro 200)

SUMMARY:
This study investigates clinical outcome and imaging outcome parameters after intraarticular injection of steroids, platelet-rich-plasma (prp), hyaluronic acid or placebo in patients with early osteoarthritis of the knee joint.

DETAILED DESCRIPTION:
Osteoarthritis of the knee joint is a very common disease in middle aged and elderly patients. This study evaluates the efficiency of different commonly used substances for intraarticular, non-operative treatment in early stages of this disease.

120 patients receive an fluoroscopic guided injection in the knee joint: 30 patients get injection with steroids 30 patients get injection with prp 30 patients get injection with hyaluronic acid 30 patients get injection with placebo (iopamiro contrast media)

Primary outcome: - clinical outcome (pain using numeric rating scale)

* Magnetic Resonance imaging (cartilage defects etc.)

ELIGIBILITY:
Inclusion criteria:

* gonarthritis Kellgren 1,2,3 with symptoms
* german speaking
* informed consent

Exclusion criteria:

-age under 18, gonarthritis, Kellgren 4, anticoagulation therapy, known inflammatory disease or infection, cardiovascular disease NYHA IV, immunosuppression, contraindication for MRI, pregnancy, no informed consent, NSAR 3 days before injection, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-02; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Pain assessment | up to 24 months after injection
  numeric rating scale (NRS) and WOMAC
Magnetic Resonance imaging | up to 12 months after injection
  cartilage volume (ml)
Magnetic Resonance imaging | up to 12 months after injection
  T2-values in cartilage (mean Signal +/- Standard Deviation) in subregions

SECONDARY OUTCOMES:
WOMAC score (stiffness, difficulty) | up to 24 months after injection
  Clinical outcome
Tegner Activity Scale | up to 24 months after injection
  Clinical outcome
Knee mobility and thigh circumference | 3 month after injection
  Clinical assessment, comparison to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Rosskopf, MD, Principal Investigator — Radiology University Hospital Balgrist
Locations (1):
- University Hospital Balgrist, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tschopp M, Pfirrmann CWA, Brunner F, Fucentese SF, Galley J, Stern C, Sutter R, Catanzaro S, Kuhne N, Rosskopf AB. Morphological and Quantitative Parametric MRI Follow-up of Cartilage Changes Before and After Intra-articular Injection Therapy in Patients With Mild to Moderate Knee Osteoarthritis: A Randomized, Placebo-Controlled Trial. Invest Radiol. 2024 Sep 1;59(9):646-655. doi: 10.1097/RLI.0000000000001067. Epub 2024 Feb 28. PMID 38421679
- [Derived] Tschopp M, Pfirrmann CWA, Fucentese SF, Brunner F, Catanzaro S, Kuhne N, Zwyssig I, Sutter R, Gotschi T, Tanadini M, Rosskopf AB. A Randomized Trial of Intra-articular Injection Therapy for Knee Osteoarthritis. Invest Radiol. 2023 May 1;58(5):355-362. doi: 10.1097/RLI.0000000000000942. Epub 2022 Dec 27. PMID 36728848